CLINICAL TRIAL: NCT05408572
Title: A Phase 1, Randomized, Adaptive-Design, Dose-Escalation Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of SON-1010 (IL12-FHAB) in Healthy Adults
Brief Title: Study of SON-1010 (IL12-FHAB) in Healthy Adults
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Sonnet BioTherapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: SB102
Record Dates: First submitted 2022-06-01; First posted 2022-06-07 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Healthy Adult

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Single Dose Level 1 (Experimental): 6 healthy adults dosed with SON-1010 (Level 1) + 2 healthy adults dosed with Placebo
  Interventions: Biological: SON-1010 (IL12-FHAB)
- Single Dose Level 2 (Experimental): 6 healthy adults dosed with SON-1010 (Level 2) + 2 healthy adults dosed with Placebo
  Interventions: Biological: SON-1010 (IL12-FHAB)
- Single Dose Level 3 (Experimental): 6 healthy adults dosed with SON-1010 (Level 3) + 2 healthy adults dosed with Placebo
  Interventions: Biological: SON-1010 (IL12-FHAB)
- Single Dose Level 4 (Experimental): 6 healthy adults dosed with SON-1010 (Level 4) + 2 healthy adults dosed with Placebo
  Interventions: Biological: SON-1010 (IL12-FHAB)
- Single Dose Level 5 (Experimental): 6 healthy adults dosed with SON-1010 (Level 5) + 2 healthy adults dosed with Placebo
  Interventions: Biological: SON-1010 (IL12-FHAB)

INTERVENTIONS:
Biological: SON-1010 (IL12-FHAB) — SON-1010 is a single-chain human IL-12 cytokine linked to a single-chain variable region known as the FHAB.

SUMMARY:
SB102 is a randomized, double-blind, single center, placebo-controlled study in healthy adults starting with sentinel participants at each dose level to carefully assess the safety, tolerability, PK, and PD of SON-1010.

DETAILED DESCRIPTION:
This is a study of SON-1010, a single-chain human Interleukin-12 (IL12) cytokine linked to a single-chain variable region (scFv) antibody fragment, known as the fully human albumin binding domain (FHAB). The albumin binding domain moiety of SON-1010 attaches to albumin in the bloodstream, resulting in significantly enhanced drug PK properties, potentially lower risk than IL12 alone, and a broader therapeutic index. Healthy volunteers will be assessed with single ascending doses of SON-1010. The design comprises up to 5 separate dosing cohorts, with a total of 8 participants (minimum of 7) in each cohort randomized to receive either SON-1010 (6 participants) or placebo (2 participants), for up to 40 participants.

ELIGIBILITY:
Inclusion Criteria

* Participants must be medically healthy based on medical history, physical examination, and clinical laboratory testing.
* Participants must be between 18 to 54 years of age, inclusive at the time of the informed consent.
* May only be limited users of nicotine-containing products, including e-cigarettes, for at least 3 continuous months before the first dose of SON-1010, as confirmed by cotinine testing at screening and check-in (day -1). Social smoking is allowed up to 5 cigarettes per week as long as the participant is willing to abstain during confinement and the cotinine test is negative at check in. One repeat test is permitted at screening.
* Must have negative drug/alcohol testing at screening and check-in (day -1). Screening drug/alcohol testing may be repeated once if deemed appropriate.
* Must have vital signs (after sitting for at least 5 minutes) within the following ranges at screening and check-in (day -1):

  * Systolic blood pressure (BP), 90 to 140 mmHg, inclusive
  * Diastolic BP, 40 to 90 mmHg, inclusive
  * Heart rate (HR) >50 to ≤100 beats per minute
* Must weigh >50 kg and ≤100 kg and have body mass index (BMI) ≥18 and ≤32 kg/m2 at screening.
* Must have normal laboratory function by day -1 (note that the screening safety laboratory assessment may be repeated once to confirm the initial result and trending), defined as:

  * Creatinine level ≤ upper limit of normal (ULN) for age
  * Alanine aminotransferase (ALT) ≤ ULN
  * Total bilirubin ≤ ULN (unless participant has Grade 1 bilirubin elevation due to Gilbert's disease or a similar syndrome involving slow conjugation of bilirubin and direct bilirubin is <35%)
  * Albumin > lower limit of normal (LLN)
  * Coagulation International Normalized Ratio (INR) < 1.5
* Females of childbearing potential, <1-year postmenopause who are not permanently sterile, must have a negative serum pregnancy test (beta-human chorionic gonadotropin [β-HCG]) at day -1, and agree to abstinence or use 2 highly effective methods of birth control for 30 days before the study, during the study, and for 30 days after the last dose of study intervention. Females who are not of childbearing potential (have had a hysterectomy, bilateral oophorectomy, or are ≥ 1-year postmenopause) do not need to use any contraception Nonchildbearing potential is defined as surgically sterile or postmenopausal (defined as 12 months of spontaneous amenorrhea). A follicle stimulating hormone (FSH) level >40 IU/L at screening will confirm postmenopausal status. If a participant is not sexually active, but becomes active, then she and her male partner must use 2 methods of adequate contraception.
* Males and their female partners must use a highly effective method of birth control if female partner(s) is of childbearing potential and must not donate sperm during the study and for 90 days after the last dose of study intervention. Contraception guidance is described in the protocol.
* Willing and able to provide signed informed consent as described in the protocol which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.
* Must be able to communicate well with Investigator and/or study site personnel and to comply with the requirements of the entire study.

Exclusion Criteria

* Concurrent conditions that could interfere with safety and/or tolerability measurements.
* Known history of allergy to any component of study intervention.
* History of severe allergic/anaphylactic reaction.
* Pregnancy and/or lactation
* Receipt of any plasma-, protein-, or antibody-based therapeutic agents (e.g., growth hormones or monoclonal antibodies) within 3 months before the first dose of study intervention. Note: Influenza and COVID-19 vaccines will be allowed if administered more than 14 days before the first dose of study intervention.
* Receipt of any investigational agent or treatment within 30 days or 5 half-lives, whichever is longer, before the first dose of study intervention.
* Any active infection, including COVID-19, as determined by the currently applicable standard before study intervention.
* Any acute noninfectious illness within 30 days before day 1.
* Diagnosis of or positive screening result for active COVID-19, hepatitis B surface antigen (HbsAg), hepatitis C virus antibody (HCVAb), or human immunodeficiency virus (HIV)-1 or HIV-2 antibody.
* Unable or unwilling to cooperate with the Investigator for any reason.
* History of any clinically relevant or chronic psychiatric, renal, hepatic, cardiovascular, pancreatic, neurologic, hematologic, or gastrointestinal disease (e.g., inflammatory bowel disease) or current clinically significant liver function test results. Mild anxiety and depression may be acceptable at the investigator's discretion.
* Evidence of any surgical or medical condition that, in the judgment of the Investigator, might interfere with the absorption, distribution, metabolism, or excretion of study intervention. History of cholecystectomy is acceptable.
* Presence of clinically significant electrocardiogram (ECG) finding (confirmed upon repeat testing) that may interfere with any aspect of study conduct or interpretation of results, as follows:

  * QT interval corrected for HR according to Fridericia's formula (QTcF) > 450 in males or > 470 msec in females at screening or check-in (day -1).
  * Other ECG abnormalities clinically relevant in the judgment of the Investigator.
* Use of any prescription or over-the-counter medications (apart from standard doses of analgesics), herbal products (e.g., St. John's Wort, garlic supplements, milk thistle), topical or inhaled steroids, or supplements/vitamins within 7 days before the first dose of SON-1010 and for the duration of the study, except for those approved by the Investigator and Sponsor (e.g., oral contraceptives, hormone replacement therapy).
* Recent use of systemic steroids within 14 days of enrollment, except for physiologic doses for steroid replacement. Limited doses of systemic steroids (e.g., in patients with exacerbation of reactive airway disease) must have been completed at least 10 days before enrollment.
* Use of biotin (i.e. Vitamin B7) or supplemental biotin higher than the daily adequate intake of 30 μg (FDA 2019). Patients who switch from a high dose to a dose of 30 μg/day or less are eligible.
* History of alcohol or substance abuse within 6 months before the first dose of SON-1010 per the criteria in the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-V).
* History of any major surgery within 3 months before the first dose of study intervention.
* Donation or receipt of blood or blood product within 3 months before the first dose of SON-1010 and for the duration of the study.

Ages: 18 Years to 54 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2022-07-27 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-05-17 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of SON-1010 as a single-ascending dose (SAD) in healthy adults. | Study Duration - Week 1 on Day 1, 2, 3 ,4, 5. Follow-Up on Day 8, 10, 12, 15, 22, 29
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0

SECONDARY OUTCOMES:
Serum and urine concentrations of SON-1010 will be determined at various time points | Study Duration - Week 1 on Day 1, 2, 3 ,4, 5. Follow-Up on Day 8, 10, 12, 15, 22, 29
  Concentration vs time of SON-1010 will be measured using blood & urine samples taken at various time points on study
Effect of SON-1010 on Serum cytokine levels | Study Duration - Week 1 on Day 1, 2, 3 ,4, 5. Follow-Up on Day 8, 10, 12, 15, 22, 29
  Concentration of serum level of IL-2, IL-6, IL-10 will be measured using blood samples taken at various time points on study
Evaluation of SON-1010 immunogenicity | Study Duration - Week 1 on Day 1, 2, 3 ,4, 5. Follow-Up on Day 8, 10, 12, 15, 22, 29
  Evaluate the immunogenicity of SON-1010 by measuring the number of patients developing anti-SON-1010 antibodies

CONTACTS AND LOCATIONS:
Overall Officials: Richard Kenney, MD, Study Director — Sonnet BioTherapeutics
Locations (1):
- Nucleus Network Pty Ltd, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kenney RT, Cini JK, Dexter S, DaFonseca M, Bingham J, Kuan I, Chawla SP, Polasek TM, Lickliter J, Ryan PJ. A phase I trial of SON-1010, a tumor-targeted, interleukin-12-linked, albumin-binding cytokine, shows favorable pharmacokinetics, pharmacodynamics, and safety in healthy volunteers. Front Immunol. 2024 Feb 29;15:1362775. doi: 10.3389/fimmu.2024.1362775. eCollection 2024. PMID 38487528